CLINICAL TRIAL: NCT06482047
Title: Rejuvenating the Brain and Boosting Executive Function With Exercise Intervention
Brief Title: Boosting Executive Function With Brain Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liye Zou (Other)
Responsible Party: Sponsor-Investigator, Liye Zou, Professor, Shenzhen University
Organization: Shenzhen University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ShenzhenUExerciseIntervention
Record Dates: First submitted 2024-01-03; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: The study used a within-participant cross-over design with pre-and post-test comparisons. Participants completed the three following experimental conditions in pseudo-counterbalanced (cannot be completely counterbalanced given that an odd number of participants - hence, was pseudo-counterbalanced) order (odd number of participants) with at least a 7-day washout period between conditions: (i) 115-minute uninterrupted sitting [control]; (ii) 50-minute sitting + 15-minute moderate-intensity cycling + 50-minute sitting [experimental condition 1]; (iii) 50-minute sitting + 15-minute vigorous-intensity cycling + 50-minute sitting [experimental condition 2]. A familiarization session was completed about three days before the experiment started, during which participants were familiarized with the cognitive assessment and cycling protocols.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate-intensity cycling (Experimental): Moderate-intensity cycling on Ergoline Ergoselect 100
  Interventions: Behavioral: Moderate-intensity cycling; Behavioral: Uninterrupted sitting
- Vigorous-intensity cycling (Experimental): Vigorous-intensity cycling on Ergoline Ergoselect 100
  Interventions: Behavioral: Vigorous-intensity cycling; Behavioral: Uninterrupted sitting
- Uninterrupted sitting (Experimental): Uninterrupted sitting in a quiet room
  Interventions: Behavioral: Uninterrupted sitting

INTERVENTIONS:
Behavioral: Moderate-intensity cycling — Moderate-intensity cycling on Ergoline Ergoselect 100
  Arms: Moderate-intensity cycling
Behavioral: Vigorous-intensity cycling — Vigorous-intensity cycling on Ergoline Ergoselect 100
  Arms: Vigorous-intensity cycling
Behavioral: Uninterrupted sitting — Uninterrupted sitting in a quiet room

SUMMARY:
The goal of this study is to explore the impact of a 15-minute exercise break on brain function and cognitive performance in a simulated classroom setting. The main questions it aims to answer are:

1. How do short exercise breaks affect executive function in college students?
2. What changes occur in brain connectivity and microcirculation after these exercise breaks? Participants were college students who engaged in sessions of continuous sitting or sitting interspersed with exercise. The study used cognitive tasks and brain imaging techniques to measure the effects. The findings reveal improvements in cognitive performance and brain function, suggesting that short exercise breaks are beneficial in educational contexts.

ELIGIBILITY:
Inclusion Criteria:

-right-handed (how was handedness assessed; i.e., "What hand do you write with?") with normal or corrected-to-normal vision and normal color vision

Exclusion Criteria:

-reported a history of cardiovascular, metabolic, gastrointestinal, neurological, or psychiatric disorders, medical conditions requiring medical care, substance addiction, strict diets (e.g., low- carbohydrate and Mediterranean diet), pregnancy, or lactation.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-02 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 3 weeks
  This primary outcome measure is assessed by the modified dual-task Stroop paradigm.
Retinal Vessel Diameter | 3 weeks
  Retinal Vessel Diameter is assessed by the fully automated fundus camera.
Brain Connectivity | 3 weeks
  Brain connectivity is assessed by the NIRSport2 device

CONTACTS AND LOCATIONS:
Locations (1):
- Body-Brain-Mind Laboratory, School of Psychology, Shenzhen University, Shenzhen, China